CLINICAL TRIAL: NCT06221709
Title: Continuous Radiofrequency in Hip Osteoarthritis Pain: A Protocol of a Randomized Clinical Trial
Brief Title: Continuous Radiofrequency in Hip Osteoarthritis Pain: A Randomized Clinical Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: Sarah Network of Rehabilitation Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: f3356f
Record Dates: First submitted 2024-01-14; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-09

CONDITIONS: Hip Osteoarthritis; Hip Pain Chronic
Keywords: denervation; Radiofrequency ablation
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants will be blinded to which group they will be allocated, as well as data assessors, who will not have contact with participants on the day of the procedure. In order to avoid differentiating the number of perforations needed to perform each procedure, all patients will receive the same bandage (Opsite®) in the anterior region of the hip, with instruction to remove it only the day after the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): This group will be submitted to an intraarticular infiltration of corticosteroid + anesthetic.
  Interventions: Procedure: Intraarticular Infiltration ( Control group)
- CRF group (Experimental): This group will be submitted to radiofrequency for sensitive hip branches from the Femoral and Obturator nerves followed by an intraarticular infiltration of corticosteroid + anesthetic similar to the control group.
  Interventions: Procedure: Conventional Radiofrequency (CRF group)

INTERVENTIONS:
Procedure: Conventional Radiofrequency (CRF group) — Radiofrequency will be performed with a 22-gauge CRF cannula, 10/15 cm long, 10mm curved active tip, at 90º for 90 seconds, introduced in the anteroposterior and lateromedial directions, to reach the teardrop landmark. Denervation of the articular branches of the Obturator Nerve will be performed in 2 cycles, starting lateral to the lateral edge of the obturator foramen, followed by a point approximately 1cm lateral to the first point. Next, the cannula will be repositioned in a more cranial location, parallel to the superolateral edge of the acetabular dome, to reach the sensory branches of the Femoral Nerve, performing 3 cycles at the 01, 12, and 11 o'clock positions. All lesions will be preceded by motor stimulation at 2,5V and cycles will be followed by the infusion of 2ml of 1% ropivacaine. After concluding the procedure, hip intraarticular infiltration will be performed as described for the control group.
  Other Names: Radioablation
  Arms: CRF group
Procedure: Intraarticular Infiltration ( Control group) — For the control group (IA), an epidural anesthesia needle (22G spinal needle) will be used, positioned anteroposteriorly towards the central portion of the femoral neck, which will be introduced until transfixion of the anterior hip capsule through tactile sensitivity. After checking the correct positioning with the use of fluoroscopy and infusion of 3 ml of 50% diluted iodinated contrast, an infusion of 4 ml of 1% Ropivacaine and 80mg of methylprednisolone 40mg/ml will be done.
  Arms: Control Group

SUMMARY:
This will be a prospective, single-center, double-blinded, randomized study designed to compare the efficacy of the intraarticular injection of a corticosteroid and the Conventional Radiofrequency (CRF) of the anterior sensory branches to the hip in controlling pain and improving function related to hip osteoarthritis.

DETAILED DESCRIPTION:
Procedures will be performed in the surgical block of Hospital SARAH, Brasília unit, using an aseptic technique.

All participants will undergo sedation or general anesthesia using a laryngeal mask airway, according to the preference of the anesthetist in the room. The procedure will be performed with the participant positioned in dorsal decubitus, on a radiolucent table, with a small pillow below the knees to promote a slight flexion of 10 to 20 degrees of the hips, leading to relaxation of the joint capsule.

The surgeon will be positioned at the side of the surgical table, facing the affected hip, with the scoping device on the contralateral side, aligned at 90 degrees with the patient, allowing the visualization of anteroposterior images of the affected hip.

For the control group (IAI), a 22G spinal needle will be used, positioned in the anteroposterior direction towards the central portion of the femoral neck, which will be introduced until it trespasses the anterior hip capsule through tactile sensitivity. After verifying the correct positioning with the use of fluoroscopy and infusion of 3 milliliters (ml) of iodinated contrast diluted at 50% (Iomeron® 300, Patheon Italia S.p.A. Ferentino - Italy), an infiltration of 4 ml of 1% Ropivacaine (Ropi®, Cristália, Itapira - São Paulo, Brazil) and 80mg of methylprednisolone 40mg/ml (Predi-Medrol®, União Química, Brasília - Federal District, Brazil) will be performed, totalizing 6 ml of solution.

In the intervention group (IA + CRF), radiofrequency ablation will be performed with the aid of a 22-gauge cannula (Diros Technology Inc, Markham, Ontario, Canada), 10 or 15 cm long, with a 10-mm curved active tip, at a temperature of 90º for 90 seconds. The cannula will be introduced in the region just above the tip of the greater trochanter, lateral to a descending line originating in the anterior superior iliac spine (ASIS), and directed to the medial border of the patella (ASIS - patella). Its introduction will take place in the anteroposterior and lateromedial direction, to reach the region lateral to the anatomical reference known as the teardrop, with an angle of about 20 to 30 craniocaudal degrees about a transverse line on the axis of the thigh. The denervation of the articular branches of the Obturator Nerve (NO) will be performed in 2 cycles, at a temperature of 90 degrees for 90 seconds, starting lateral to the lateral edge of the obturator foramen and inferior to the teardrop, with subsequent repositioning of the cannula about 1 cm lateral to the first point. Both lesions will be preceded by motor stimulation at 2.5 volts (V) to exclude motor branches within the range of action of the active tip followed by the infusion of 2ml of 1% ropivacaine. Then, the cannula will be repositioned in a more cranial location, 2 to 3 cm lateral to the ASIS-patella line, parallel to the superolateral edge of the acetabular dome, to reach the sensory branches of the Femoral Nerve (NF), performing three cycles (from medial to lateral) at the 01, 12, and 11 o'clock positions. The most medial lesion will be preceded by motor stimulation at 2.5 V to exclude motor branches within the active tip's range of action. All three cycles will be followed by 2 ml of 1% ropivacaine infusion. After completion of radiofrequency ablation, IAI of the hip will follow as described for the control group above.

ELIGIBILITY:
Inclusion Criteria:

* Individuals ≥ 18 years of age, with symptomatic unilateral hip osteoarthritis, grades II and III according to the Kellgreen and Lawrance classification, hip pain for more than six months (medial, anterior, anterolateral, and/or lateral region) will be included.

Exclusion Criteria:

* Individuals with radiculopathy and ipsilateral irradiation, osteonecrosis of the femoral head, previous arthroplasty on the hip to be studied or surgical scar that could lead to changes in the anatomy of the hip, cases of high dislocation of the hip, pain exclusively in the posterior region, symptomatic ipsilateral knee osteoarthritis, intra-articular infiltration of corticosteroids or hyaluronic acid in the hip for less than six months, patients with neurological diseases, peripheral neuropathy or psychiatric diseases, use of a pacemaker or Prothrombin Activity Time (INR) > 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (WOMAC) | Baseline to 24 weeks ± 1 week.
  The Western Ontario and McMaster Universities (WOMAC) is a self-administered health status measure and consists of 24 items divided into three domains, which are pain (5 questions), stiffness (2 questions), and physical function (17 questions), validated to patients with hip or knee osteoarthritis, available in a 5-point Likert scale, ranging from 0 to 96 points.This questionnaire is translated and validated in portuguese.

SECONDARY OUTCOMES:
Change in Pain Visual Analogue Scale | Baseline, 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week
  The pain visual analogue scale (VAS) is a unidimensional measure of pain intensity, in a continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme, "no pain" (score 0) and " worst pain ever" (score 100).
Pain Medication Intake | Baseline, 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  To evaluate pain medication we will use a scale ranging from 0 to 4 (0= no medication; 0 = no medication; 1= use of dipyrone or paracetamol; 2= use of NSAIDs; 3= use of opiate derivatives; 4= routinely scheduled opiate derivatives), considering the last 48 hours.
Change in Hip muscles Isometric Peak Force | Baseline, 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  To examine isometric muscle force, a Lafayette Manual Muscle Testing System Model-01165 (Lafayette Instrument Company, Lafayette IN, USA) will be used to access Peak Force of hip flexors, abductors, adductors and extensors.
Change in Hip muscles Average Force | Baseline, 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  To examine isometric muscle force, a Lafayette Manual Muscle Testing System Model-01165 (Lafayette Instrument Company, Lafayette IN, USA) will be used to access Average Force of hip flexors, abductors, adductors and extensors. We will also determine intra and inter-rater reliability for isometric force of hip flexors, abductors, adductors and extensors.
Change in Global Satisfaction | Time Frame: 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week
  To evaluate participant satisfaction, we will use 5 points Likert Scale, ranging from 0 to 4 (0= none _ no good at all, ineffective intervention; 1= poor _ some effect but unsatisfactory; 2= fair _ reasonable effect but could be better; 3= good _ satisfactory effect with occasional episodes of pain or stiffness; 4= excellent _ ideal response, virtually pain-free).
Incidence of Adverse Effects | 1 week, 12 weeks ± 1 week and 24 weeks ± 1 week.
  To examine the incidence of adverse effects, a questionnaire will be apply to investigate the occurrence of: Hematoma, paresthesia, weakness, worsening of pain, worsening of function or any other adverse effect that participants attribute to the procedure performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Rede Sarah Hospitais de Reabilitação, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Non-identified data will be provided for peer revision in an Open database to allow verification of conclusions as well as inclusion in metanalysis studies.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available at the moment of publication of the final paper.
Access Criteria: Open access.

REFERENCES:
- [Background] Learmonth ID, Young C, Rorabeck C. The operation of the century: total hip replacement. Lancet. 2007 Oct 27;370(9597):1508-19. doi: 10.1016/S0140-6736(07)60457-7. PMID 17964352
- [Background] Singh JA, Schleck C, Harmsen S, Lewallen D. Clinically important improvement thresholds for Harris Hip Score and its ability to predict revision risk after primary total hip arthroplasty. BMC Musculoskelet Disord. 2016 Jun 10;17:256. doi: 10.1186/s12891-016-1106-8. PMID 27286675
- [Background] Pulik L, Romaniuk K, Jaskiewicz K, Wojtynski P, Legosz P, Maldyk P. An update on joint-specific outcome measures in total hip replacement. Reumatologia. 2020;58(2):107-115. doi: 10.5114/reum.2020.95366. Epub 2020 Apr 30. PMID 32476684
- [Background] Chye CL, Liang CL, Lu K, Chen YW, Liliang PC. Pulsed radiofrequency treatment of articular branches of femoral and obturator nerves for chronic hip pain. Clin Interv Aging. 2015 Mar 16;10:569-74. doi: 10.2147/CIA.S79961. eCollection 2015. PMID 25834413
- [Background] McCabe PS, Maricar N, Parkes MJ, Felson DT, O'Neill TW. The efficacy of intra-articular steroids in hip osteoarthritis: a systematic review. Osteoarthritis Cartilage. 2016 Sep;24(9):1509-17. doi: 10.1016/j.joca.2016.04.018. Epub 2016 Apr 30. PMID 27143362
- [Background] Corbett KL, Losina E, Nti AA, Prokopetz JJ, Katz JN. Population-based rates of revision of primary total hip arthroplasty: a systematic review. PLoS One. 2010 Oct 20;5(10):e13520. doi: 10.1371/journal.pone.0013520. PMID 20976011
- [Background] Ajrawat P, Radomski L, Bhatia A, Peng P, Nath N, Gandhi R. Radiofrequency Procedures for the Treatment of Symptomatic Knee Osteoarthritis: A Systematic Review. Pain Med. 2020 Feb 1;21(2):333-348. doi: 10.1093/pm/pnz241. PMID 31578561
- [Background] Roberts SL, Stout A, Dreyfuss P. Review of Knee Joint Innervation: Implications for Diagnostic Blocks and Radiofrequency Ablation. Pain Med. 2020 May 1;21(5):922-938. doi: 10.1093/pm/pnz189. PMID 31407791
- [Background] Gofeld M, Restrepo-Garces CE, Theodore BR, Faclier G. Pulsed radiofrequency of suprascapular nerve for chronic shoulder pain: a randomized double-blind active placebo-controlled study. Pain Pract. 2013 Feb;13(2):96-103. doi: 10.1111/j.1533-2500.2012.00560.x. Epub 2012 May 4. PMID 22554345
- [Background] Kawaguchi M, Hashizume K, Iwata T, Furuya H. Percutaneous radiofrequency lesioning of sensory branches of the obturator and femoral nerves for the treatment of hip joint pain. Reg Anesth Pain Med. 2001 Nov-Dec;26(6):576-81. doi: 10.1053/rapm.2001.26679. PMID 11707799
- [Background] Kumar P, Hoydonckx Y, Bhatia A. A Review of Current Denervation Techniques for Chronic Hip Pain: Anatomical and Technical Considerations. Curr Pain Headache Rep. 2019 May 1;23(6):38. doi: 10.1007/s11916-019-0775-z. PMID 31044316
- [Background] Bhatia A, Hoydonckx Y, Peng P, Cohen SP. Radiofrequency Procedures to Relieve Chronic Hip Pain: An Evidence-Based Narrative Review. Reg Anesth Pain Med. 2018 Jan;43(1):72-83. doi: 10.1097/AAP.0000000000000694. PMID 29140960
- [Background] Rivera F, Mariconda C, Annaratone G. Percutaneous radiofrequency denervation in patients with contraindications for total hip arthroplasty. Orthopedics. 2012 Mar 7;35(3):e302-5. doi: 10.3928/01477447-20120222-19. PMID 22385437
- [Background] Vanaclocha-Vanaclocha V, Sáiz-Sapena N, Herrera JM, Rivera-Paz M, Verdú-López F, Renovell-Ferrer P, et al. Cronicon EC ORTHOPAEDICS Clinical Study Percutaneous Radiofrequency Denervation in the Treatment of Hip Pain Secondary to Osteoarthritis. n.d.
- [Background] Chan A-W, Tetzlaff JM, Altman DG, Laupacis A, Gøtzsche PC, Krleža-Jeric K, et al. SPIRIT 2013 Statement: Defining Standard Protocol Items for Clinical Trials DEVELOPMENT OF THE SPIRIT 2013 STATEMENT. vol. 158. 2013.
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Kohn MD, Sassoon AA, Fernando ND. Classifications in Brief: Kellgren-Lawrence Classification of Osteoarthritis. Clin Orthop Relat Res. 2016 Aug;474(8):1886-93. doi: 10.1007/s11999-016-4732-4. Epub 2016 Feb 12. No abstract available. PMID 26872913
- [Background] Bang H, Flaherty SP, Kolahi J, Park J. Blinding assessment in clinical trials: A review of statistical methods and a proposal of blinding assessment protocol. Clin Res Regul Aff 2010;27:42-51. https://doi.org/10.3109/10601331003777444.
- [Background] James KE, Bloch DA, Lee KK, Kraemer HC, Fuller RK. An index for assessing blindness in a multi-centre clinical trial: disulfiram for alcohol cessation--a VA cooperative study. Stat Med. 1996 Jul 15;15(13):1421-34. doi: 10.1002/(SICI)1097-0258(19960715)15:133.0.CO;2-H. PMID 8841652
- [Background] Fernandes M. MARCUS IVANOVITH FERNANDES TRADUÇÃO E VALIDAÇÃO DO QUESTIONÁRIO DE QUALIDADE DE VIDA ESPECÍFICO PARA OSTEOARTROSE WOMAC (Western Ontario and McMaster Universities) PARA A LÍNGUA PORTUGUESA. São Paulo : 2002.
- [Background] Garbuz DS, Xu M, Sayre EC. Patients' outcome after total hip arthroplasty: a comparison between the Western Ontario and McMaster Universities index and the Oxford 12-item hip score. J Arthroplasty. 2006 Oct;21(7):998-1004. doi: 10.1016/j.arth.2006.01.014. PMID 17027542
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Leão MG de S, Martins Neta GP, Coutinho LI, da Silva TM, Ferreira YMC, Dias WRV. Análise comparativa da dor em pacientes submetidos à artroplastia total do joelho em relação aos níveis pressóricos do torniquete pneumático. Rev Bras Ortop (Sao Paulo) 2016;51:672-9. https://doi.org/10.1016/j.rbo.2016.02.002.
- [Background] DeLoach LJ, Higgins MS, Caplan AB, Stiff JL. The visual analog scale in the immediate postoperative period: intrasubject variability and correlation with a numeric scale. Anesth Analg. 1998 Jan;86(1):102-6. doi: 10.1097/00000539-199801000-00020. PMID 9428860
- [Background] Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi: 10.1002/acr.20543. No abstract available. PMID 22588748
- [Background] Lane NE, Hochberg MC, Nevitt MC, Simon LS, Nelson AE, Doherty M, Henrotin Y, Flechsenhar K. OARSI Clinical Trials Recommendations: Design and conduct of clinical trials for hip osteoarthritis. Osteoarthritis Cartilage. 2015 May;23(5):761-71. doi: 10.1016/j.joca.2015.03.006. PMID 25952347
- [Background] Mentiplay BF, Perraton LG, Bower KJ, Adair B, Pua YH, Williams GP, McGaw R, Clark RA. Assessment of Lower Limb Muscle Strength and Power Using Hand-Held and Fixed Dynamometry: A Reliability and Validity Study. PLoS One. 2015 Oct 28;10(10):e0140822. doi: 10.1371/journal.pone.0140822. eCollection 2015. PMID 26509265
- [Background] Chamorro C, Armijo-Olivo S, De la Fuente C, Fuentes J, Javier Chirosa L. Absolute Reliability and Concurrent Validity of Hand Held Dynamometry and Isokinetic Dynamometry in the Hip, Knee and Ankle Joint: Systematic Review and Meta-analysis. Open Med (Wars). 2017 Oct 17;12:359-375. doi: 10.1515/med-2017-0052. eCollection 2017. PMID 29071305
- [Background] Walter SD, Eliasziw M, Donner A. Sample size and optimal designs for reliability studies. Stat Med. 1998 Jan 15;17(1):101-10. doi: 10.1002/(sici)1097-0258(19980115)17:13.0.co;2-e. PMID 9463853
- [Background] Tinnirello A, Todeschini M, Pezzola D, Barbieri S. Pulsed Radiofrequency Application on Femoral and Obturator Nerves for Hip Joint Pain: Retrospective Analysis with 12-Month Follow-up Results. Pain Physician. 2018 Jul;21(4):407-414. PMID 30045597